CLINICAL TRIAL: NCT03324581
Title: A Phase 2, Multicenter, Randomized, Double-blind, Active- and Placebo-controlled Trial of the Safety and Efficacy of OPC-64005 in the Treatment of Adult Attention-deficit/Hyperactivity Disorder
Brief Title: The Safety and Efficacy of OPC-64005 in the Treatment of Adult Attention-deficit/Hyperactivity Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 277-201-00001
Record Dates: First submitted 2017-10-25; First posted 2017-10-27 (Actual); Results first posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-09

CONDITIONS: Adult Attention Deficit Hyperactivity Disorder
Keywords: ADHD; ADD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OPC-64005 (Experimental): During the titration period, participants received OPC-64005 two 10 milligram (mg) tablets, and one OPC-64005-matching placebo tablet along with two atomoxetine-matching placebo capsules, orally, once daily (QD), from Day 1 up to Day 4. During the treatment period, participants received OPC-64005 three 10 mg tablets, and two atomoxetine-matching placebo capsules, orally, QD, from Day 5 up to Day 56. The dose was reduced to 20 mg if the 30 mg dose in the treatment period was not tolerable.
  Interventions: Drug: OPC-64005; Drug: Placebo
- Atomoxetine (Active Comparator): During the titration period, participants received atomoxetine one 40 mg capsule and one atomoxetine-matching placebo capsule along with three OPC-64005-matching placebo tablets, orally, QD, from Day 1 up to Day 4.
  During the treatment period, participants received two atomoxetine 40 mg capsules and three OPC-64005-matching placebo tablets, orally, QD, from Day 5 up to Day 56. The dose was reduced to 40 mg if the 80 mg dose in the treatment period was not tolerable.
  Interventions: Drug: Atomoxetine; Drug: Placebo
- Placebo (Placebo Comparator): Participants received three OPC-64005-matching placebo tablets and two atomoxetine-matching placebo capsules, orally, QD, from Day 1 up to Day 56.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OPC-64005 — OPC-64005 film coated tablets
  Arms: OPC-64005
Drug: Atomoxetine — Atomoxetine gelatin capsules
  Arms: Atomoxetine
Drug: Placebo — OPC-64005-matching placebo film coated tablets and atomoxetine-matching placebo gelatin capsules

SUMMARY:
A trial to assess the safety and efficacy of OPC-64005 in the treatment of adult attention-deficit/hyperactivity disorder.

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, active- and placebo-controlled, parallel-design trial.

ELIGIBILITY:
Inclusion Criteria (Screening):

* Male and female participants 18 to 55 years of age, inclusive, at the time of informed consent.
* Participants with a primary Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) diagnosis of ADHD (including predominantly inattentive presentation, hyperactive presentation, and combined presentations) as confirmed by the Adult ADHD Clinical Diagnostic Scale (ACDS) v 1.2.
* Participants willing to discontinue all prohibited psychotropic medication starting from the time of signing the informed consent and up to the 30 (+ 2)-day follow-up period.

Exclusion Criteria:

* Participants with a history of inadequate response or suboptimal tolerability to atomoxetine.
* Participants who report allergies (lifetime treatment history) to stimulant or nonstimulant ADHD medications.
* Participants with other DSM-5 disorders including psychosis (current or lifetime), bipolar disorder (current or lifetime), current major depressive disorder, or current panic disorder; or another psychiatric diagnosis that the investigator believes is primary or that will confound efficacy or safety assessments of the trail or interfere with participation in the trial otherwise.
* Participants with a clinically significant current DSM-5 diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal, histrionic, narcissistic, avoidant, obsessive compulsive, or dependent personality disorders.
* Participants who currently have clinically significant dermatological, neurological, hepatic, renal, metabolic, hematological, immunological, cardiovascular, pulmonary, or gastrointestinal disorders such as any history of myocardial infarction, congestive heart failure, HIV (human immunodeficiency virus) seropositive status/acquired immunodeficiency syndrome, or active or chronic hepatitis B or C.
* Participants with a history of obstructive sleep apnea.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 239 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Southern California Research, LLC, Beverly Hills, California
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Artemis Institute for Clinical Research, San Marcos, California
  - MCB Clinical Research Centers, LLC, Colorado Springs, Colorado
  - Meridien Research, Bradenton, Florida
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - Behavioral Clinical Research, Inc., North Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Clinical Neuroscience Solutions Inc., Orlando, Florida
  - iResearch Atlanta, Decatur, Georgia
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Psychiatric Associates, Overland Park, Kansas
  - Premier Psychiatric Research Institute, LLC, Lincoln, Nebraska
  - Center for Psychiatry and Behavioral Medicine Inc., Las Vegas, Nevada
  - Eastside Comprehensive Medical Center, LLC., New York, New York
  - The Medical Research Network, LLC, New York, New York
  - IPS Research Company, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigators, Inc., Portland, Oregon
  - Oregon Center for Clinical Investigators, Inc., Salem, Oregon
  - BTC of Lincoln, Lincoln, Rhode Island
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Aspen Clinical Research, Orem, Utah
  - Neuropsychiatric Associates, Woodstock, Vermont

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 26 sites in the United States from 09 November 2017 to 31 October 2018.
Pre-assignment Details: Participants with adult attention deficit hyperactivity disorder (ADHD) were randomized in 1:1:1 ratio into the titration period to receive OPC-64005, atomoxetine, and placebo. This was followed by the treatment period wherein the dose was escalated based on tolerability.
Period: Overall Study
Arm/Group | OPC-64005 | Atomoxetine | Placebo
Started | 77 | 80 | 82
Completed | 38 | 44 | 57
Not Completed | 39 | 36 | 25
Not completed — Adverse Event | 18 | 11 | 7
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Lost to Follow-up | 5 | 3 | 6
Not completed — Non-Compliance With Investigational Medicinal Product (IMP) | 2 | 2 | 0
Not completed — Physician Decision | 0 | 1 | 2
Not completed — Protocol Deviation | 8 | 9 | 4
Not completed — Withdrawal by Subject | 6 | 8 | 6
Not completed — Day 56 Visit was 15 Days Out of the Visit Window | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Analysis Set included all participants who were randomized in the trial.
Groups:
- OPC-64005: During the titration period, participants received OPC-64005 two 10 mg tablets, and one OPC-64005-matching placebo tablet along with two atomoxetine-matching placebo capsules, orally, QD, from Day 1 up to Day 4. During the treatment period, participants received OPC-64005 three 10 mg tablets, and two atomoxetine-matching placebo capsules, orally, QD, from Day 5 up to Day 56. The dose was reduced to 20 mg if the 30 mg dose in the treatment period was not tolerable.
- Total: Total of all reporting groups
Arm/Group | OPC-64005 | Atomoxetine | Placebo | Total
Number analyzed (Participants) | 77 | 80 | 82 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (8.6) | 35.1 (8.8) | 34.6 (9.3) | 35.1 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 46 | 42 | 127
  Male | 38 | 34 | 40 | 112
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 58 | 60 | 64 | 182
  Race: Black or African American | 7 | 15 | 12 | 34
  Race: American Indian or Alaska Native | 3 | 2 | 2 | 7
  Race: Asian | 2 | 1 | 2 | 5
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Race: Other | 7 | 1 | 1 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 21 | 18 | 17 | 56
  Ethnicity: Not Hispanic or Latino | 55 | 62 | 65 | 182
  Ethnicity: Unknown | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Conners' Adult ADHD Rating Scales-Observer: Screening Version (CAARS-O:SV) 18-item ADHD Symptoms Total Score at Day 56
Description: The investigator-administered CAARS-O:SV consists of 18 items based on the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5). It includes a 9-item inattentive symptom subscale and a 9-item hyperactive and impulsive symptoms subscale. Each item is rated on a scale of 0 to 3 where 0=not at all, never; 1=just a little, once a while; 2=pretty much, often; and 3=very much, very frequently. The score for each subscale can range from 0 to 27. The total score is the sum of individual scores and can range from 0 to 54. Higher scores indicate worsening of symptoms. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Day 56
Population: Full Analysis Set (FAS) included all randomized participants who took at least one dose of IMP and had a Baseline and at least one post randomization evaluation for the CAARS-O:SV ADHD Symptoms total score (18-items). Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OPC-64005 | Atomoxetine | Placebo
Number analyzed (Participants) | 76 | 74 | 77
score on a scale
  Baseline | 40.71 (6.99) | 41.59 (6.66) | 40.51 (7.10)
  Change at Day 56: number analyzed (Participants) | 42 | 50 | 59
  Change at Day 56 | -19.4 (17.79) | -20.2 (13.24) | -10.3 (13.52)
Statistical Analysis 1: Comparison: OPC-64005 vs Atomoxetine; Test type: Superiority; p = 0.7554, Mixed-effect Model Repeated Measures — The change from baseline in CAARS-O:SV was analyzed using a Mixed-effect Model Repeated Measures (MMRM) methodology with the unstructured variance covariance matrix; It included fixed class-effect terms: treatment,trial site,visit week, interaction term: treatment by visit week, Baseline CAARS-O:SV as a covariate; Difference = 0.81, 95% CI 2-sided [-4.30 to 5.92]
Statistical Analysis 2: Comparison: OPC-64005 vs Placebo; Test type: Superiority; p = 0.0101, Mixed-effect Model Repeated Measures — The change from baseline in CAARS-O:SV was analyzed using a MMRM methodology with the unstructured variance covariance matrix; [statistical method as in outcome 1, analysis 1]; Difference = -6.61, 95% CI 2-sided [-11.6 to -1.60]
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority; p = 0.0033, Mixed-effect Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference = -7.42, 95% CI 2-sided [-12.3 to -2.50]

2. Other Pre Specified Outcome: Change From Baseline in CAARS-O:SV 18-item Score on Days 7, 14, 21, 28, 42, and 56
Description: The investigator-administered CAARS-O:SV consists of 18 items based on the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria. It includes a 9-item inattentive symptom subscale and a 9- item hyperactive and impulsive symptoms subscale. Each item is rated on a scale of 0 to 3 where 0=not at all, never; 1=just a little, once a while; 2=pretty much, often; and 3=very much, very frequently. The score for each subscale can range from 0 to 27. The total score is the sum of individual scores and can range from 0 to 54. Higher scores indicate worsening of symptoms. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Days 7, 14, 21, 28, 42, and 56
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Change From Baseline in Adult ADHD Investigator Symptom Rating Scale (AISRS) With Adult Prompts Score on Day 28 and Day 56
Description: The AISRS consists of 18-items derived from DSM-IV criteria for ADHD symptoms. The AISRS total score is the sum of the 9-item inattentive symptoms subscale and 9-item hyperactive and impulsive symptoms subscale. Each item is scored as follows: 0=none, 1=mild, 2=moderate, and 3=severe. The score for each subscale can range from 0 to 27. The total score can range from 0 to 54. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Days 28 and 56
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Score on Days 7, 14, 21, 28, 42, and 56
Description: The CGI-S evaluates the severity of individual symptoms and treatment response in participants with mental disorders. It is a 7-point scale that that requires the clinician to rate the severity of the participant's illness at the time of assessment as 0=not assessed, 1=normal, not at all ill, 2=borderline mentally ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill, 7=among the most extremely ill participants. The score 0=not assessed was set to missing. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Days 7, 14, 21, 28, 42, and 56
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Clinical Global Impression-Improvement (CGI-I) Score on Days 7, 14, 21, 28, 42, and 56
Description: The CGI-I is a 7-point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to a Baseline state at the beginning of the intervention and rated as: 0=not assessed, 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse. The score of 0 =not assessed was set to missing. Lower scores indicate improvement.
Time Frame: Baseline, Days 7, 14, 21, 28, 42, and 56
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change From Baseline in Conners' Adult ADHD Rating Scales-Self-Report: Screening Version (CAARS-S:SV) 18-item Total Score on Days 7, 14, 21, 28, 42, and 56
Description: The CAARS-S:SV comprises of 30 items to measure symptoms for ADHD in adults but was limited to the 18 DSM-5 criteria relevant items for this trial. The 18-item ADHD Symptoms total score is the sum of the 9-item inattentive symptoms subscale and the 9-item hyperactive and impulsive symptoms subscale. Each item is rated on a scale of 0 to 3 where 0=not at all, never; 1=just a little, once a while; 2=pretty much, often; and 3=very much, very frequently. The score for each subscale can range from 0 to 27. Total score can range from 0 to 54. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Days 7, 14, 21, 28, 42, and 56
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change From Baseline in Adult ADHD Quality of Life Scale (AAQoL) Total Score on Day 28 and Day 56
Description: The AAQoL is a validated, 29-item instrument for measuring the impact of ADHD symptoms on quality of life. The scale assesses 4 distinct functional domains based on the following subscales: life productivity (11 items), psychological health (6 items), life outlook (7 items), and relationships (5 items). Scores for individual items range from 1=never/not at all to 5=extremely/very often. Total and subscale scores were computed by (1) reversing scores for all items except the seven items in the Life Outlook subscale; (2) transforming all item scores to a 0-100 point scale (1=0; 2=25; 3=50; 4=75; 5=100); and (3) summing item scores and dividing by the item count to generate subscale and total scores. Higher scores indicate a greater impact.
Time Frame: Baseline, Days 28, and 56
Reporting Status: Not Posted

8. Other Pre Specified Outcome: OPC-64005 Potential for Abuse Liability and Dependence as Assessed by the Drug Effects Questionnaire (DEQ) Score
Description: The DEQ was used to assess the potential for abuse of OPC-64005. It is a 5-item questionnaire completed by the participant that includes the following questions: 1. Do you feel a drug effect right now? 2. Are you high right now? 3. Do you dislike any of the effects you are feeling right now? 4. Do you like any of the effects you are feeling right now? 5. would you like more of the drug you took, right now? Each item is rated on a 100-point scale of 1 (not at all) to 100 (extremely). 100 represents the highest score for that subjective state, and the higher the score, the worse the outcome.
Time Frame: Baseline, Days 7, 14, 21, 28, 42, and 56
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days post last dose of study drug (Up to approximately 12 months)
Description: Safety Analysis Set included all participants who were randomized and administered at least 1 dose of IMP during the trial.
Arm/Group | OPC-64005 | Atomoxetine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/79 | 0/82
Serious Adverse Events (participants affected / at risk) | 1/77 | 0/79 | 0/82
Other Adverse Events (participants affected / at risk) | 61/77 | 59/79 | 38/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-64005 (N=77) | Atomoxetine (N=79) | Placebo (N=82)
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-64005 (N=77) | Atomoxetine (N=79) | Placebo (N=82)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0
Goitre (Endocrine disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Blepharitis (Eye disorders) | 0 | 0 | 1
Mydriasis (Eye disorders) | 2 | 0 | 0
Vision blurred (Eye disorders) | 1 | 3 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1
Change of bowel habit (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 5 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 15 | 9 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 2 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 14 | 20 | 2
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Chest discomfort (General disorders) | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 7 | 12 | 4
Feeling abnormal (General disorders) | 1 | 1 | 0
Feeling jittery (General disorders) | 0 | 2 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1
Temperature intolerance (General disorders) | 0 | 1 | 0
Thirst (General disorders) | 3 | 1 | 0
Body tinea (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 4 | 1 | 2
Pharyngitis (Infections and infestations) | 0 | 2 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 3
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 2
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 2 | 0
Heart rate increased (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 13 | 12 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 6 | 6 | 2
Dizziness postural (Nervous system disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 6 | 6 | 3
Hypersomnia (Nervous system disorders) | 1 | 0 | 0
Nystagmus (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 3 | 0
Poor quality sleep (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0
Sedation (Nervous system disorders) | 4 | 3 | 0
Somnolence (Nervous system disorders) | 2 | 5 | 4
Tension headache (Nervous system disorders) | 1 | 1 | 2
Tremor (Nervous system disorders) | 1 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 0
Apathy (Psychiatric disorders) | 2 | 0 | 1
Bruxism (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Depersonalisation/derealisation disorder (Psychiatric disorders) | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1
Derealisation (Psychiatric disorders) | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 2 | 0 | 1
Disturbance in sexual arousal (Psychiatric disorders) | 0 | 0 | 1
Euphoric mood (Psychiatric disorders) | 0 | 0 | 1
Illusion (Psychiatric disorders) | 0 | 0 | 1
Initial insomnia (Psychiatric disorders) | 0 | 3 | 1
Insomnia (Psychiatric disorders) | 6 | 4 | 2
Irritability (Psychiatric disorders) | 1 | 4 | 4
Libido decreased (Psychiatric disorders) | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 1
Middle insomnia (Psychiatric disorders) | 3 | 2 | 2
Nightmare (Psychiatric disorders) | 0 | 2 | 0
Orgasm abnormal (Psychiatric disorders) | 2 | 0 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0
Staring (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 2 | 0 | 0
Tearfulness (Psychiatric disorders) | 0 | 1 | 0
Terminal insomnia (Psychiatric disorders) | 2 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 1
Urinary hesitation (Renal and urinary disorders) | 2 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Ejaculation delayed (Reproductive system and breast disorders) | 2 | 0 | 0
Ejaculation disorder (Reproductive system and breast disorders) | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 6 | 3 | 0
Genital burning sensation (Reproductive system and breast disorders) | 1 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Yawning (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 5 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Piloerection (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 3 | 0
Vascular pain (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Study Protocol (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/81/NCT03324581/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT03324581/SAP_001.pdf